CLINICAL TRIAL: NCT02473276
Title: Two Dose Neuraxial Morphine for Prevention of Postdural Puncture Headache
Brief Title: 2 Dose Neuraxial Morphine for Prevention of PDPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Montefiore Medical Center (Other); Rutgers University (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Richard M. Smiley, Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAP4755
Record Dates: First submitted 2015-06-03; First posted 2015-06-16 (Estimated); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EPID PFM (Active Comparator): The group "EPID PFM" will receive 3 mg (6 ml) of preservative-free morphine, followed by 3 ml of sterile normal saline, to be administered through the epidural catheter.Sixteen to 24 hours after receiving the first study drug, the patient will then receive the identical study drug (for a total of two doses).
  Interventions: Drug: Morphine; Drug: Sterile normal saline
- EPID SAL (Sham Comparator): The placebo group, "EPID NS", will receive 6 ml of sterile normal saline via the epidural catheter followed by another 3 ml NS. Sixteen to 24 hours after receiving the first study drug,the patient will then receive the identical study drug (for a total of two doses).
  Interventions: Drug: Sterile normal saline
- IT PFM (Active Comparator): The group, "IT PFM" will receive 200 micrograms (mcg) (0.4 ml) of preservative-free morphine via the intrathecal catheter, followed by a flush of the catheter with 2 ml of sterile saline.Sixteen to 24 hours after receiving the first study drug, the patient will then receive the identical study drug (for a total of two doses).
  Interventions: Drug: Morphine; Drug: Sterile normal saline
- IT SAL (Sham Comparator): The placebo group IT SAL will receive 0.4 ml and then 2 ml of sterile normal saline through the intrathecal catheter.Sixteen to 24 hours after receiving the first study drug, the patient will then receive the identical study drug (for a total of two doses).
  Interventions: Drug: Sterile normal saline

INTERVENTIONS:
Drug: Morphine — preservative free morphine given either via an epidural or intrathecal catheter
  Other Names: Duramorph
  Arms: EPID PFM; IT PFM
Drug: Sterile normal saline — sterile normal saline, given either via an epidural or intrathecal catheter
  Other Names: Saline

SUMMARY:
Neuraxial analgesia (most commonly continuous epidural or combined spinal epidural) is the most effective modality available for pain relief during labor. Accidental dural puncture (ADP) with a large bore epidural needle and the resulting post-dural puncture headache (PDPH) is one of the most significant sources of anesthesia-related morbidity in parturients.

Epidural blood patch (EBP) is the gold standard for treatment of PDPH, and although almost always effective, can result in another ADP, as well as low back pain and lower extremity pain. For this reason, effective measures to prevent PDPH when ADP occurs would be highly valuable. One small study in which 50 women were randomly allocated to receive 2 epidural injections of morphine or saline, demonstrated a beneficial effect of epidural morphine in decreasing the incidence of PDPH.

This study aims to determine the efficacy of 2 doses of neuraxial (either epidural (EPID) or intrathecal) preservative-free morphine (PFM) to prevent headache after ADP in parturients.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double blind clinical trial. Subjects will be ASA I and II women (per American Society of Anesthesiologists Physical Status Classification System or ASA) aged 18 years and older, who are known to have had ADP with an epidural needle during placement of neuraxial labor analgesia, and have either an intrathecal catheter or epidural catheter in situ. Patients will be randomized to either receive PFM or placebo (sterile normal saline (NS or SAL)).

For patients with an epidural catheter, the group "EPID PFM" will receive 3 mg (6 ml) of PFM, followed by 3 ml of sterile normal saline to be administered through the epidural catheter. The placebo group, "EPID NS", will receive 6 ml of sterile normal saline via the epidural catheter followed by another 3 ml NS. For patients with an intrathecal catheter, the group, "IT PFM" will receive 200 micrograms (mcg) (0.4 ml) of preservative-free morphine, followed by a flush of the catheter with 2 ml of sterile saline. The placebo group will receive 0.4 ml and then 2 ml of sterile normal saline through the intrathecal catheter. Sixteen to 24 hours after receiving the first study drug, patients in all groups will be visited by an investigator, and then daily thereafter during the hospital admission. They will be evaluated for the presence of headache, analgesia requirements, need for EBP and the severity of opioid side effects. As long as the patient is afebrile, has not been experiencing severe opioid side effects and the catheter is in place and intact, the patient will then receive the identical study drug (for a total of two doses). The epidural/intrathecal catheter will be removed immediately after the second administration of the study drug.

After discharge, the patient will be followed up once daily by telephone for up to a minimum of 5 days after receiving the last dose of the study drug if they remain headache free, and for a minimum of 3 days after resolution of PDPH.

Statistical Design:

This will be a prospective randomized double blind clinical trial. The primary outcome will be the incidence of PDPH at 48 hours after ADP. The primary outcome of the trial is the incidence of PDPH at 48 hours after ADP. We will consider a difference in incidence of PDPH between the placebo and treatment groups of 25 % to be significant, based on the findings of Al Metwalli et al. (Anaesthesia. 2008; 63(8):847-50), and the meta-analysis by Heesen et al. (Int J Obstet Anesth. 2013 ; 22(1):26-30).

Estimates of PDPH rate after ADP range from 50 to 85%. Our rate at Columbia University Irving Medical Center (CUIMC) for the past several years is 66% (OB Anesthesia Division QA data). For calculation of our sample size, we determined that an absolute 25% decrease in PDPH would be clinically significant (i.e., 66% to ~40%). For a power of 90% and an alpha of 0.05, this requires 83 subjects per group (2 epidural groups compared to each other, 2 spinal groups compared to each other). We are not specifically powering this for comparison of the spinal to the epidural groups, although we will likely be able to do so. We therefore, aim to recruit 100 subjects per group (for a total of 400 across all centers) assuming 10-15% of subjects may be lost because of inadvertent withdrawal of the catheter, subject withdrawal, or lost to follow up after discharge.

This is intended to be a multicenter study involving 5 academic tertiary hospitals, having >2,000 vaginal deliveries per year. Since the rate of accidental dural puncture is between 1 and 2%, we estimate we should be able to recruit 100 subjects per year. Categorical data (presence or absence of dural puncture headache, need for epidural blood patch) will be analyzed using Chi-square analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be ASA I and II women aged 18 years and older, who are known to have had accidental dural puncture with an epidural needle during placement of neuraxial labor analgesia, and have either an intrathecal catheter or epidural catheter in place.

Exclusion Criteria:

* Past history of headache syndromes- such as migraine and cluster headaches
* History of chronic pain syndromes
* Chronic opioid use
* Illicit drug use - e.g. marijuana, heroin
* Allergy to morphine
* Intrapartum or postpartum fever ≥ 38 ° C
* Coagulopathy
* Accidental removal of the epidural or intrathecal catheter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Smiley, MD, PhD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Rutgers Health University Hospital, Newark, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Montefiore Hospital, New York, New York

REFERENCES:
- [Background] Al-metwalli RR. Epidural morphine injections for prevention of post dural puncture headache. Anaesthesia. 2008 Aug;63(8):847-50. doi: 10.1111/j.1365-2044.2008.05494.x. Epub 2008 Jun 10. PMID 18547293
- [Background] Scavone BM, Wong CA, Sullivan JT, Yaghmour E, Sherwani SS, McCarthy RJ. Efficacy of a prophylactic epidural blood patch in preventing post dural puncture headache in parturients after inadvertent dural puncture. Anesthesiology. 2004 Dec;101(6):1422-7. doi: 10.1097/00000542-200412000-00024. PMID 15564951

RESULTS

PARTICIPANT FLOW:
Groups:
- EPID PFM: The group "EPID PFM" will receive 3 mg (6 ml) of preservative-free morphine, followed by 3 mL of sterile normal saline, to be administered through the epidural catheter. 16 to 24 hours after receiving the first dose, the patient will then receive 3 mg (6 ml) of preservative-free morphine (for a total of two doses).
- EPID SAL: The placebo group, "EPID NS", will receive 6 mL of sterile normal saline via the epidural catheter followed by another 3 mL sterile normal saline. 16 to 24 hours after receiving the first dose, the patient will then receive 6 mL of sterile normal saline (for a total of two doses).
- IT PFM: The group, "IT PFM" will receive 200 micrograms (mcg) (0.4 mL) of preservative-free morphine via the intrathecal catheter, followed by a flush of the catheter with 2 mL of sterile normal saline. 16 to 24 hours after receiving the first dose, the patient will then receive 200 mcg (0.4 mL) of preservative-free morphine (for a total of two doses).
- IT SAL: The placebo group IT SAL will receive 0.4 mL and then 2 mL of sterile normal saline through the intrathecal catheter. 16 to 24 hours after receiving the first dose, the patient will then receive 0.4 mL and then 2 mL of sterile normal saline (for a total of two doses).
Period: Overall Study
Arm/Group | EPID PFM | EPID SAL | IT PFM | IT SAL
Started | 8 | 10 | 11 | 15
Completed | 8 | 10 | 11 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPID PFM | EPID SAL | IT PFM | IT SAL | Total
Number analyzed (Participants) | 8 | 10 | 11 | 15 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (2.6) | 31 (5.5) | 31.1 (5.8) | 32.9 (6.3) | 32.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 11 | 15 | 44
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 8 | 7 | 18
  Not Hispanic or Latino | 8 | 6 | 3 | 7 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 5 | 9
  White | 6 | 7 | 4 | 8 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 11 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postdural Puncture Headache
Description: The primary outcome will be the incidence of postdural puncture headache at 48 hours after accidental dural puncture. This will be determined by a face to face questionnaire and the severity of headache will be rated according to a verbal rating scale (0 -10).
Time Frame: 48 hours after accidental dural puncture
Measure: Count of Participants; unit: Participants
Arm/Group | EPID PFM | EPID SAL | IT PFM | IT SAL
Number analyzed (Participants) | 8 | 10 | 11 | 15
Participants | 3 | 4 | 8 | 10

2. Secondary Outcome: Number of Participants in Need for Epidural Blood Patch
Description: A secondary outcome will be the need for epidural blood patch at 48 hours after accidental dural puncture. This will be recorded on the study data collection sheet.
Time Frame: 48 hours after accidental dural puncture
Measure: Count of Participants; unit: Participants
Arm/Group | EPID PFM | EPID SAL | IT PFM | IT SAL
Number analyzed (Participants) | 8 | 10 | 11 | 15
Participants | 2 | 2 | 5 | 7

ADVERSE EVENTS:
Time Frame: 48 hours after accidental dural puncture
Arm/Group | EPID PFM | EPID SAL | IT PFM | IT SAL
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 3/8 | 4/10 | 8/11 | 10/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EPID PFM (N=8) | EPID SAL (N=10) | IT PFM (N=11) | IT SAL (N=15)
Postdural Puncture Headache (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT02473276/Prot_SAP_000.pdf